CLINICAL TRIAL: NCT02883413
Title: An Investigation of Cognitive Remediation Therapy as an Inpatient Intervention for Adolescents With Anorexia Nervosa
Brief Title: Cognitive Remediation Therapy for Adolescents With Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: The Hilda & Preston Davis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-012624
Record Dates: First submitted 2016-08-02; First posted 2016-08-30 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Anorexia Nervosa
Keywords: Adolescents; Cognitive Flexibility; Behavioral Flexibility
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CRT +Teach the Parent (Experimental): The Teach the Parent (TtP) addition to CRT is designed to increase parental understanding of their adolescents' thinking styles. We hypothesize that by doing so, parents will be more likely to challenge eating disorder behaviors and be less likely to accommodate behavioral symptoms of the eating disorder (e.g., make something low-fat for dinner because it will be easier). In this arm, adolescents will explain what they learned during CRT and walk their parents though at least 4 tasks during each TtP session. Parents and child will not be permitted to speak about the eating disorder during these sessions. TtP sessions will occur 3-4 times during hospitalization and will be guided by the adolescent.
  Interventions: Behavioral: CRT + Teach the Parent
- CRT + Family Fun Time (Active Comparator): In order to assess for any non-specific effects of spending non-eating disorder driven time with family, adolescents in the CRT+ Contact Control condition will be asked to spend 3-4 sessions with their parents engaging in fun activities (games, coloring, trivia). We refer to this condition as CRT + Family Fun Time (CRT+FFT). Adolescents will be asked to complete a series of fun tasks (some standardized, some are choice driven) with their parents. During these sessions, they will not be permitted to discuss CRT or the eating disorder.
  Interventions: Behavioral: CRT + Contact Control
- Treatment as Usual (TAU) (No Intervention): Adolescents in this condition will not receive any additional treatment. They will have a standard hospital stay with all normal contact with health professionals.

INTERVENTIONS:
Behavioral: CRT + Teach the Parent — CRT sessions will occur for 45-60 minutes every day (excluding weekends) for 6-8 days while adolescents are in hospital. Adolescents will be given homework and asked to practice tasks each day.
  Other Names: CRT+ TtP
  Arms: CRT +Teach the Parent
Behavioral: CRT + Contact Control — Adolescents will be asked to spend 3-4 sessions with their parents engaging in fun activities (games, coloring, trivia). Adolescents will be able to choose 2 tasks from a list and be asked to engage in those tasks with their parents.
  Other Names: CRT + Family Fun Time, or CRT + FFT
  Arms: CRT + Family Fun Time

SUMMARY:
The purpose of the current study is to investigate the role of Cognitive Remediation Therapy (CRT) as a pre-treatment intervention for adolescents who are hospitalized for Anorexia Nervosa (AN). The primary aims are to determine if CRT can result in greater treatment engagement post-discharge, increased rate of weight gain post-discharge, reduction in symptom accommodation, and increased behavioral flexibility in adolescents and parents.

DETAILED DESCRIPTION:
Anorexia Nervosa (AN) is a severe psychiatric condition; the hallmark features are low body weight and difficulties gaining weight. We are in need of new methods to jump start treatment, while targeting relevant processes in individuals with AN.

Study Design:

This is a randomized controlled trial looking to address these concerns, with a focus on three distinct aims:

1. To evaluate the feasibility and acceptability (by patients and staff) of CRT in a medical hospitalization setting.
2. Compare the impact of CRT to CRT + Teach the Parent on adolescent treatment engagement post-discharge, rate of weight gain post-discharge, and reduction of symptom accommodation.
3. To evaluate cognitive and behavioral flexibility 6 months post-discharge.

Setting/Participants:

Participants will be 60 adolescents with AN or subclinical AN (and their parents). Adolescents will be hospitalized for treatment of AN and intervention will occur on an inpatient basis. Follow-up will be outpatient.

Study Interventions and Measures:

The current study will investigate the impact of intensive CRT (one sessions/day) delivered during in hospital for medical stabilization. Shortly after admission to hospital, adolescents will be randomly assigned to one of the following conditions: Treatment as usual (TAU), CRT+Contact Control (known as "Family Fun Time" or FFT) and CRT + Teach the Parent. Psychosocial, neurocognitive, and behavioral measures will be collected throughout the study. Follow-up will continue for 6 months post-discharge.

Description of Investigational Intervention:

CRT is an adjunctive intervention focusing on the development of meta-cognition: Teaching individuals to think about how they think. It involves presenting individuals with a variety of tasks requiring increasingly complex mental abilities. These include sorting tasks where rules change, geometric figures, illusions, reversing sequences of numbers and letters, and finding various routes on a map.

CRT's focus is mainly on process, instead outcome, and has three main goals:

1. Improve brain function by exercising and increasing connections in the brain
2. Encourage individuals to think about their thinking style
3. Encourage individuals and families to spend time away from thinking about the eating disorder

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent is between 12-18 years of age and living at home, parent or primary caregiver willing to participate in condition they are randomized into
2. Adolescent meets diagnostic criteria of anorexia nervosa (either restricting or binge/purge subtype), or sub threshold AN according to Diagnostic and Statistical Manual-5 criteria
3. Consent of all family members who will be participating in treatment
4. Adolescent is not currently receiving outpatient treatment for the eating disorder

Exclusion Criteria:

1. Caregiver or adolescent with a co-morbid diagnosis of psychotic disorder, substance dependence, substance abuse, or bi-polar disorder
2. caregiver or adolescent with diagnosis of mental retardation, pervasive developmental disorder, or autism spectrum disorder
3. Adolescent with a diagnosis of feeding or eating concerns not elsewhere classified with the primary symptoms of bingeing and purging, binging without compensatory behaviors or spitting food or with restricting patterns
4. Adolescent with diagnosis of avoidant/restrictive food intake disorder.
5. Adolescent or caregiver with acute suicide risk.
6. Concurrent psychosocial treatment for another condition
7. Adolescent or parent not fluent in English

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08; Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Change in adolescent treatment engagement via questionnaire | Baseline to 3 months post baseline
  The Motivational Stages of Change for Adolescents Recovering from an Eating Disorder (MSCARED) is a questionnaire designed to assess readiness to change among individuals with eating disorders. It is administered via interview, discussing motivation, actions that qualify for making changes, and asking what stage of change the patient is in. The patient then checks off those actions they are doing that contribute to their recovery from a provided checklist.

SECONDARY OUTCOMES:
Change in adolescent cognitive flexibility via questionnaire | Baseline to 6 months post baseline
  The Cognitive Flexibility Scale (CFS) is a 12-item self report measure that assesses 3 different components: cognitive flexibility, rigidity and communication flexibility. Scores for each question range from 1-6 (strongly disagree - strongly agree). Scores on cognitive flexibility are positively related to communication flexibility and negatively related to rigidity. Scores on communication flexibility are also negatively related to rigidity.
Change in parental symptom accommodation, via questionnaire | Baseline to 3 months post baseline
  The Accommodation and Enabling Scale for Eating Disorders (AESED) is a 39-item measure that gathers information about the enabling behaviors that family members with a child who has an eating disorder engage in. It contains three subscales: avoidance and modifying routine, meal ritual, and control of the family.

CONTACTS AND LOCATIONS:
Overall Officials: C. Alix Timko, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Timko CA, Fitzpatrick KK, Goulazian T, Kirby D, Parks E, Morrow L, Scharko AM, Peebles R. Conducting a Pilot Randomized Controlled Trial on a Medical Inpatient Unit Utilizing Cognitive Remediation Therapy for Adolescents with Restrictive Eating Disorders: Protocol Updates and Reflections on Feasibility. J Clin Psychol Med Settings. 2020 Jun;27(2):226-234. doi: 10.1007/s10880-020-09704-w. PMID 32052249
- [Derived] Timko CA, Goulazian TJ, Fitzpatrick KK, Rodriguez D. Cognitive remediation therapy (CRT) as a pretreatment intervention for adolescents with anorexia nervosa during medical hospitalization: a pilot randomized controlled trial protocol. Pilot Feasibility Stud. 2018 Jun 25;4:87. doi: 10.1186/s40814-018-0277-5. eCollection 2018. PMID 29983992